CLINICAL TRIAL: NCT03853330
Title: Erector Spinae Plane Block Versus Thoracic Epidural Analgesia in Patients With Multiple Fracture Ribs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Hamed, Ass. Prof. in Anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Analgesia for Fracture Ribs
Record Dates: First submitted 2019-02-20; First posted 2019-02-25 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Fracture; Rib, Multiple
MeSH Terms: conditions — Fractures, Bone | interventions — Ultrasonography; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: prospective, double-blinded controlled trial; both the patient and data collector is unaware of the study nature
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic Epidural Analgesia group (Active Comparator): 25 patients will receive ultrasound-guided thoracic epidural analgesia for multiple fracture ribs at the level of T8 with 7.5-12 ml of Bupivacaine HCl Inj 0.25% as a loading dose followed by catheter insertion and infusion of Bupivacaine Hydrochloride, 0.125%-0.9% Injectable Solution at 5-7 ml/h. For breakthrough pain bolus of Bupivacaine Hydrochloride, 0.125%-0.9% Injectable Solution 5-10 ml can be used.
  Interventions: Device: Ultrasound; Drug: Bupivacaine HCl Inj 0.25%; Drug: Bupivacaine Hydrochloride, 0.125%-0.9% Injectable Solution
- Erector spinae plane block group (Active Comparator): 25 patients will receive ultrasound-guided ESP block for multiple fracture ribs at the level from T1 to T5 with 7.5-12 ml of Bupivacaine HCl Inj 0.25% as a loading dose followed by catheter insertion and infusion of Bupivacaine Hydrochloride, 0.125%-0.9% Injectable Solution at 5-7 ml/h. For breakthrough pain bolus of Bupivacaine Hydrochloride, 0.125%-0.9% Injectable Solution 5-10 ml can be used.
  Interventions: Device: Ultrasound; Drug: Bupivacaine HCl Inj 0.25%; Drug: Bupivacaine Hydrochloride, 0.125%-0.9% Injectable Solution

INTERVENTIONS:
Device: Ultrasound — Ultrasound-guided Thoracic Epidural Analgesia and Erector spinae plane block.
Drug: Bupivacaine HCl Inj 0.25% — Bupivacaine HCl Inj 0.25% will be used in both blocks by the same dose of 7.5-12 ml
Drug: Bupivacaine Hydrochloride, 0.125%-0.9% Injectable Solution — infusion of Bupivacaine Hydrochloride, 0.125%-0.9% Injectable Solution at 5-7 ml/h will be used in both blocks and also for breakthrough pain after both blocks as a bolus of 5-10 ml.

SUMMARY:
To assess the analgesic and respiratory effect of continuous Erector Spinae Plane block versus Thoracic Epidural in patients with multiple fracture ribs.

DETAILED DESCRIPTION:
Erector spinae plane (ESP) block is a recently described technique which may be an alternative to Paravertebral block (PVB) for providing thoracic analgesia. It involves injection of local anesthetic into the fascial plane deep to erector spinae muscle. ESP is a more superficial block with a better defined end-point injection between the bony transverse process and erector spinae muscle. A more superficial ultrasound-guided block will be faster to perform and less painful for the patient. ESP does not have the same risk of pneumothorax as PVB.

Epidural analgesia has become the standard of care. Although thoracic epidurals provide excellent analgesia for the management of rib fractures, they are limited to a certain population due to patient factors and side-effects. Many trauma patients have other injuries which contraindicate the use of epidurals, or which prevent positioning for insertion. There are disadvantages to thoracic epidural analgesia. They are technically challenging to insert, with a risk of dural puncture or spinal cord injury. Adverse effects include hypotension, and if opioids used, urinary retention and pruritus. Patients can develop a motor block and are unable to mobilize with an epidural in situ.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple fracture ribs.

Exclusion Criteria:

* Patient refusal.
* Patients with pre-existing infection at the block site.
* Coagulopathy.
* Allergy to local anesthetics.
* Pre-existing neurological deficits.
* Psychiatric illness.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Pain score (verbal numeric rating scale) as the median VNRS at rest and cough | up to 24 hours
  All patients will be assessed for pain score using the 11 points verbal numeric rating scale (VNRS), where zero equals no pain and 10 equals the worst pain imaginable. This assessment will be done before the block and after the block by 60 minutes and then every 6 hours up to 24 hours.

SECONDARY OUTCOMES:
Pulmonary function test | up to 24 hours
  Pulmonary function test will be done before the block, 60 minutes after the block and then every 6 hours up to 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt